CLINICAL TRIAL: NCT05743868
Title: Metabolic Heterogeneity Underlying Hypertriglyceridemia: Hepatic Triglyceride Biosynthesis in Humans With Different Insulin Resistance Phenotypes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Amsterdam UMC (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Vatner 012523; NL83166.018.22 (Other: Amsterdam UMC); R01DK124272 (NIH)
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Insulin Resistance; Hypertriglyceridemia
MeSH Terms: conditions — Insulin Resistance; Hypertriglyceridemia

STUDY DESIGN:
Intervention Model Description: Glucose tolerance, skeletal muscle/whole-body insulin sensitivity and adipose tissue insulin sensitivity will be evaluated prior to intervention. Plasma deuterium will be allowed to wash out over several weeks, and the 2nd deuterated water study will be performed.
  Randomized crossover within group design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IR participants with standardized dinner (Experimental): Participants with global IR and tissue-specific IR. Participants with global IR (in both skeletal muscle and adipose tissue) and tissue-specific IR (in adipose tissue). Glucose tolerance, skeletal muscle/whole-body insulin sensitivity and adipose tissue insulin sensitivity will be evaluated prior to intervention.
  Contribution of DNL to hepatic VLDL will be measured using a deuterated water drink, to be ingested prior to the standardized dinner. Blood will be drawn the following morning for the measurement of deuterium incorporation into triglycerides. Plasma deuterium will be allowed to wash out over several weeks, and the 2nd deuterated water study will be performed.
  Interventions: Behavioral: Standardized Dinner
- IR participants with standardized dinner and premeal exercise (Experimental): Participants with global IR and tissue-specific IR. Participants with global IR (in both skeletal muscle and adipose tissue) and tissue-specific IR (in adipose tissue). Glucose tolerance, skeletal muscle/whole-body insulin sensitivity and adipose tissue insulin sensitivity will be evaluated prior to intervention.
  DNL will be assessed in all participants after a single day with short bouts of premeal exercise with a standardized dinner.
  Contribution of DNL to hepatic VLDL will be measured using a deuterated water drink, to be ingested prior to the standardized dinner. Blood will be drawn the following morning for the measurement of deuterium incorporation into triglycerides. Plasma deuterium will be allowed to wash out over several weeks, and the 2nd deuterated water study will be performed.
  Interventions: Behavioral: Standardized Dinner; Behavioral: Premeal exercise

INTERVENTIONS:
Behavioral: Standardized Dinner — De novo lipogenesis (DNL) will be assessed in all participants with a standardized dinner
Behavioral: Premeal exercise — DNL will be assessed in all participants with short bouts of premeal exercise with a standardized dinner
  Arms: IR participants with standardized dinner and premeal exercise

SUMMARY:
The focus of this cross-sectional study is to determine the effects of tissue-specific (adipose tissue or muscle) vs global (combined) insulin resistance (IR) on hepatic triglyceride biosynthesis in humans, and to determine differential effects of an acute exercise intervention on hepatic triglyceride biosynthesis in these groups.

DETAILED DESCRIPTION:
Hypothesis: Patients who primarily have muscle IR will have a greater percentage of lipids derived from de novo lipogenesis (DNL) than patients with combined muscle and adipose IR, and these subjects will respond more robustly to the effects of premeal exercise.

With this study, the investigators will demonstrate that the mechanisms that drive triglyceride overproduction in insulin-resistant humans are dependent on which tissues are insulin resistant. To this end, investigators will determine whether subjects with muscle insulin resistance and adipose tissue insulin resistance utilize different mechanisms of triglyceride biosynthesis to assemble hepatic very low density lipoprotein (VLDL), as compared with individuals with muscle insulin resistance but relative adipose tissue insulin sensitivity. Additionally, investigators will see if adipose tissue insulin sensitivity predicts exercise responsiveness of hepatic triglyceride production.

Main study parameters/endpoints: Difference in %DNL between subjects with global vs muscle-only insulin resistance as well as the differential effects of premeal exercise on %DNL in these groups.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Overweight, defined as BMI 25-30 kg/m2
* Modest hypertriglyceridemia, defined as fasting plasma triglycerides 1.5-3.0mM
* High risk of insulin resistance, defined as fasting plasma insulin >64pM
* Stable weight for at least 3mo prior to participation

Exclusion Criteria:

* Active or chronic liver disease, kidney disease, congestive heart failure, unstable angina, history of acute cardiovascular events within 6mo of screening, history of seizures or syncope, or an active infection requiring antimicrobial therapy;
* Use of insulin, thiazolidinediones, SGLT2 inhibitors, or sulfonylureas;
* Use of fibrates, omega 3 (fish oil), niacin, or PCSK9 antagonists;
* Use of systemic glucocorticoids within 60d prior to participation;
* Hematocrit <35%;
* Pregnancy of breastfeeding;
* Active tobacco use, excessive alcohol intake (>14U/wk), or history of drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Effect of tissue-specific insulin resistance on contribution of DNL to plasma triglyceride | Baseline
  The amount of de novo lipogenesis (DNL) in VLDL-triglycerides after a standard meal will be measured in plasma from whole blood. Relationship between DNL and 1) whole body (skeletal muscle) insulin resistance and 2) white adipose tissue insulin resistance will be assessed individually.
Change in DNL in VLDL-triglycerides after a standard meal compared to a standard meal with premeal exercise. | study visit 1 and study visit 2, up to 8 weeks
  The amount of de novo lipogenesis (DNL) in VLDL-triglycerides after a standard meal vs after a standard meal with premeal exercise will be measured in plasma from whole blood.

SECONDARY OUTCOMES:
Change in plasma triglycerides after a standard meal compared to a standard meal with premeal exercise | study visit 1 and study visit 2, up to 8 weeks
  Plasma triglycerides will be measured under both conditions.
Baseline plasma triglycerides | baseline
  Plasma triglycerides will be measured at the screening visit to determine eligibility for the study
Adipose insulin sensitivity | Baseline
  Both nonesterified fatty acids and insulin will be measured in the plasma at baseline to calculate Adipo-IR, a measure of adipose tissue insulin sensitivity.
Skeletal muscle/whole-body insulin sensitivity assessed by oral glucose tolerance test (OGTT) | Baseline
  Matsuda index will be used to evaluate whole body physiological insulin sensitivity from the data obtained by OGTT. Insulin sensitivity as calculated by the Matsuda index: [10,000 / √glucose minute 0 x insulin minute 0) (mean glucose (OGTT) x mean insulin OGTT)]. A higher result indicates less IR.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Vatner, MD, PhD, Principal Investigator — Yale University
Locations (1):
- AMC Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
By reasonable request, PI can be reached by email, and individual participant data (OGTT results, fasting plasma data, DNL data) will be provided electronically.
Time Frame: Data will be available when data collection ends until 36 months after publication.